CLINICAL TRIAL: NCT04406688
Title: Prediction of Acute Kidney Injury in Patients With COVID-19 Associated Acute Respiratory Distress Syndrome
Brief Title: Prediction of Acute Kidney Injury in Patients With COVID-19
Status: Completed | Type: Observational
Sponsor: University Hospital Muenster (Other)
Responsible Party: Sponsor
Other Study IDs: 04-AnIt-20
Record Dates: First submitted 2020-05-18; First posted 2020-05-28 (Actual); Last update posted 2022-11-07 (Actual); Status verified 2022-11

CONDITIONS: Acute Kidney Injury; COVID-19; ARDS
Keywords: biomarker
MeSH Terms: conditions — Acute Kidney Injury; COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — EDTA plasma, urine
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The two biomarkers determined in urine, "Tissue Inhibitor of Metalloproteinases 2 (TIMP-2)" and "Insulin-like Growth Factor-Binding Protein 7 (IGFBP7)", can indicate the occurrence of Acute kidney injury (AKI) in cardiac surgery and critically ill patients at an early stage. However, no data are available whether these parameters can also predict the occurrence of AKI in the context of COVID-19 infection. An early prediction of AKI can be helpful for the optimisation of therapeutic management to improve patient outcome and for the triage of patients.

The aim of this observational study is to evaluate whether the biomarker [TIMP- 2]*[IGFBP7] can predict the occurrence of AKI in critically ill patients suffering from SARS-CoV2 associated acute respiratory distress syndrome.

DETAILED DESCRIPTION:
Severe Acute Respiratory Syndrome Coronavirus 2 (SARS-CoV-2) is rapidly spreading around the world. The current outbreak of infections with SARS-CoV-2 is termed Coronavirus Disease 2019 (COVID-19). Two other coronavirus infections, SARS in 2002-2003 and Middle East Respiratory Syndrome (MERS) in 2012, both caused severe respiratory syndrome in humans. All 3 of these emerging infectious diseases are caused by β-coronaviruses.

Although COVID-19 primarily affects the lungs and may cause severe hypoxemia, other organs including the GI tract, heart and kidney are affected. Acute kidney injury secondary to COVID-19 (COV-AKI) is reported to occur in about 15-25% of patients hospitalized with COVID-19 infection. The majority of AKI cases are mild to moderate with renal replacement requirement in about 25%. However, AKI was much more common in non-survivors (>50%). Although kidney failure appears to occur late in the course, patients may begin to develop AKI within the first 3 days of hospitalization. Similar to AKI in other settings,3 COV-AKI is likely to be of variable etiology. Thus, there may be a long window for treatment.

The two cell-cycle arrest markers, tissue inhibitor of metalloproteinases-2 (TIMP-2) and insulin-like growth-factor binding protein 7 (IGFBP7), have been shown to early predict the occurrence of AKI in cardiac surgical and critically ill patients. However, there is no data available whether (TIMP-2)*(IGFBP7) can predict the occurrence of AKI in the COVID19 setting. Early prediction of AKI may be valuable to optimize therapeutic management in order to improve patient's outcome and might be helpful to triage patients.

The goal of this observational trial is to evaluate whether (TIMP-2)*(IGFBP7) early predicts the occurrence of AKI in critically ill patients with SARS-CoV2 associated ARDS.

ELIGIBILITY:
Inclusion Criteria:

1. Moderate or severe ARDS according to the Berlin definition
2. SARS-CoV2 positive test
3. Age ≥ 18 years
4. Informed consent

Exclusion Criteria:

1. Pre-existing AKI
2. Severe CKD with eGFR<20ml/min
3. Chronic dialysis dependency
4. Kidney transplant within the last 12 months
5. Pregnancy, breastfeeding
6. Persons with any kind of dependency on the investigator or employed by the sponsor or investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Primary care clinic
Sampling Method: Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2020-06-22 (Actual); Primary Completion 2021-12-30 (Actual); Study Completion 2022-03-31 (Actual)

PRIMARY OUTCOMES:
Occurence of acute kidney injury (AKI) | within 7 days after beginning of moderate or severe ARDS
  Occurence of moderate or severe AKI

SECONDARY OUTCOMES:
Occurence of transient and persistent AKI | within 7 days after beginning of moderate or severe ARDS
Occurence of Renal replacement therapy during hospital stay | up to 4 weeks after beginning of moderate or severe ARDS
Duration of renal replacement therapy | up to 4 weeks after beginning of moderate or severe ARDS
Mortality | up to 4 weeks after beginning of moderate or severe ARDS
Duration of mechanical ventilation | up to 4 weeks after beginning of moderate or severe ARDS
Duration of vasopressor administration | up to 4 weeks after beginning of moderate or severe ARDS
ICU length of stay | up to 4 weeks after beginning of moderate or severe ARDS
Hospital length of stay | up to 4 weeks after beginning of moderate or severe ARDS

OTHER OUTCOMES:
Concentration of pro- and antiinflammatory mediators | within 7 days after beginning of moderate or severe ARDS
  Add-on-Analysis: Concentration of interleukin (IL) 6, IL8

CONTACTS AND LOCATIONS:
Overall Officials: Alexander Zarbock, MD, Study Chair — University Hospital Muenster, Dept. of Anesthesiology, Intensive Care Medicine and Pain Therapy
Locations (13):
- University Hospital Münster, Münster, Germany
- Italy (2):
  - Papa Giovanni XXIII Hospital, Bergamo
  - San Bortolo Hospital, Vicenza
- Portugal (2):
  - Centro Hospitalar e Universitário de Coimbra, Coimbra
  - Centro Hospitalar e Universitário do Porto, Porto
- Spain (7):
  - Hospital de la Vall d'Hebron, Barcelona
  - Hospital Germans Trias i Pujol, Barcelona
  - Hospital Sant Pau, Barcelona
  - University Hospital SAS de Jere, Jerez de la Frontera
  - Complejo Hospitalario de Navarra, Pamplona
  - Hospital Universitario Mutua Terrassa, Terrassa
  - Hospital la Fe, Valencia
- Guy's & St. Thomas Hospital, London, United Kingdom

REFERENCES:
- [Derived] Weiss R, von Groote T, Ostermann M, Lumlertgul N, Weerapolchai K, Garcia MIM, Cano JMM, Del Corral BD, Broch-Porcar MJ, Perez Carrasco M, De la Vega Sanchez A, Sousa E, Catarino A, Roig AJB, Martinez de Irujo JB, de Rosa S, de la Pena MG, Tomasa T, Brivio M, De Molina FJG, Gerss J, Kellum JA, Wempe C, Leidereiter A, Meersch M, Zarbock A. The Role of Cell Cycle Arrest Biomarkers for Predicting Acute Kidney Injury in Critically Ill COVID-19 Patients: A Multicenter, Observational Study. Crit Care Med. 2023 Aug 1;51(8):992-1000. doi: 10.1097/CCM.0000000000005853. Epub 2023 Mar 28. PMID 36975308